CLINICAL TRIAL: NCT06428708
Title: Comparison of [18F] PSMA-1007 PET/CT and Conventional Imaging in the Detection of Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: [18F] PSMA-1007 PET/CT in Metastatic Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Western University (Other)
Responsible Party: Principal Investigator, Melissa Huynh, Assistant Professor, Western University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ReDA 11465
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
Keywords: PSMA PET; Metastatic clear cell renal cell carcinoma; [18F]PSMA-1007; PSMA
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F] PSMA-1007 PET/CT (Experimental): All patients enrolled undergo a [18F] PSMA-1007 PET/CT
  Interventions: Diagnostic Test: [18F] PSMA-1007 PET/CT

INTERVENTIONS:
Diagnostic Test: [18F] PSMA-1007 PET/CT — [18F] PSMA-1007 PET/CT scan

SUMMARY:
Staging of kidney cancer is primarily achieved by computerized tomography (CT) scans or magnetic resonance imaging (MRI). If a patient is found to have limited metastatic disease, surgical removal or radiation therapy could be considered in order to control the majority of the disease. However, if metastases are more widespread, systemic (drug) therapy may be the preferred management option. The identification of additional metastatic sites using more sensitive imaging modalities therefore has the potential to alter management, and this remains an unmet need in the field. This study will investigate the utility of positron emission tomography (PET) imaging with PSMA (prostate specific membrane antigen). Kidney cancer of the clear cell subtype has demonstrated high expression of PSMA, making it a disease in which PSMA-targeted PET imaging could help to identify occult metastatic disease.

DETAILED DESCRIPTION:
This will be a single-institution prospective, open-label feasibility study involving patients ≥18 years of age with metastatic clear cell RCC who have not yet received systemic therapy. Patients with evidence of metastatic disease on conventional imaging will require histologic confirmation by biopsy. At our institution, approximately 26 new metastatic clear cell RCC (mRCC) patients are seen each year, and a previous analysis reported that 92% of 10,105 patients with mRCC in the International mRCC Database Consortium (IMDC) database were found to have clear cell histology; therefore, difficulty with recruitment into this study over a period of 2 years is not anticipated.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with histologically-proven, metastatic renal cell carcinoma (RCC)(TNM stage Tany, Nany, M1)
2. Must have baseline conventional imaging of the chest, abdomen, and pelvis with contrast-enhanced CT or MRI within 5 weeks of enrolment. Contrast is required unless the participant cannot for medical reasons (ie renal failure).

Exception: Unenhanced CT of the chest is acceptable Exception: Unenhanced MRI of abdomen and pelvis is acceptable in cases of renal failure

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Age less than 18
3. Histology does not have any clear cell component
4. Unable to lie flat for 30 minutes for the scan
5. History of prior malignancy (except non-melanoma skin cancer)
6. Unable to provide informed consent
7. Inadequate liver function
8. Systemic or radiation-based cancer treatment is needed urgently and anticipated to begin before PSMA scan can take place
9. Previously exposed to systemic or radiation cancer therapy (except radiation for skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of metastatic lesions | 5 weeks from initial baseline conventional imaging
  To identify additional metastatic lesions that may not be apparent on conventional cross-sectional imaging during the initial staging process.
Change in management | 1 month
  To determine the proportion of patients in which results from the PSMA-PET imaging changes management.

SECONDARY OUTCOMES:
Pathologic correlates | 1 month or not applicable
  To determine histopathological correlation in lesions that are biopsied or removed surgically.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Huynh, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mittlmeier LM, Unterrainer M, Rodler S, Todica A, Albert NL, Burgard C, Cyran CC, Kunz WG, Ricke J, Bartenstein P, Stief CG, Ilhan H, Staehler M. 18F-PSMA-1007 PET/CT for response assessment in patients with metastatic renal cell carcinoma undergoing tyrosine kinase or checkpoint inhibitor therapy: preliminary results. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):2031-2037. doi: 10.1007/s00259-020-05165-3. Epub 2020 Dec 28. PMID 33369689
- [Background] Giesel FL, Hadaschik B, Cardinale J, Radtke J, Vinsensia M, Lehnert W, Kesch C, Tolstov Y, Singer S, Grabe N, Duensing S, Schafer M, Neels OC, Mier W, Haberkorn U, Kopka K, Kratochwil C. F-18 labelled PSMA-1007: biodistribution, radiation dosimetry and histopathological validation of tumor lesions in prostate cancer patients. Eur J Nucl Med Mol Imaging. 2017 Apr;44(4):678-688. doi: 10.1007/s00259-016-3573-4. Epub 2016 Nov 26. PMID 27889802
- [Background] Rhee H, Blazak J, Tham CM, Ng KL, Shepherd B, Lawson M, Preston J, Vela I, Thomas P, Wood S. Pilot study: use of gallium-68 PSMA PET for detection of metastatic lesions in patients with renal tumour. EJNMMI Res. 2016 Dec;6(1):76. doi: 10.1186/s13550-016-0231-6. Epub 2016 Oct 22. PMID 27771904
- [Background] Yin Y, Campbell SP, Markowski MC, Pierorazio PM, Pomper MG, Allaf ME, Rowe SP, Gorin MA. Inconsistent Detection of Sites of Metastatic Non-Clear Cell Renal Cell Carcinoma with PSMA-Targeted [18F]DCFPyL PET/CT. Mol Imaging Biol. 2019 Jun;21(3):567-573. doi: 10.1007/s11307-018-1271-2. PMID 30218388
- [Background] Meyer AR, Carducci MA, Denmeade SR, Markowski MC, Pomper MG, Pierorazio PM, Allaf ME, Rowe SP, Gorin MA. Improved identification of patients with oligometastatic clear cell renal cell carcinoma with PSMA-targeted 18F-DCFPyL PET/CT. Ann Nucl Med. 2019 Aug;33(8):617-623. doi: 10.1007/s12149-019-01371-8. Epub 2019 May 30. PMID 31147927
- [Background] Baccala A, Sercia L, Li J, Heston W, Zhou M. Expression of prostate-specific membrane antigen in tumor-associated neovasculature of renal neoplasms. Urology. 2007 Aug;70(2):385-90. doi: 10.1016/j.urology.2007.03.025. PMID 17826525
- [Background] Chang SS, Reuter VE, Heston WD, Gaudin PB. Metastatic renal cell carcinoma neovasculature expresses prostate-specific membrane antigen. Urology. 2001 Apr;57(4):801-5. doi: 10.1016/s0090-4295(00)01094-3. PMID 11306418
- [Background] Kinoshita Y, Kuratsukuri K, Landas S, Imaida K, Rovito PM Jr, Wang CY, Haas GP. Expression of prostate-specific membrane antigen in normal and malignant human tissues. World J Surg. 2006 Apr;30(4):628-36. doi: 10.1007/s00268-005-0544-5. PMID 16555021
- [Background] Prasad V, Steffen IG, Diederichs G, Makowski MR, Wust P, Brenner W. Biodistribution of [(68)Ga]PSMA-HBED-CC in Patients with Prostate Cancer: Characterization of Uptake in Normal Organs and Tumour Lesions. Mol Imaging Biol. 2016 Jun;18(3):428-36. doi: 10.1007/s11307-016-0945-x. PMID 27038316
- [Background] Park JW, Jo MK, Lee HM. Significance of 18F-fluorodeoxyglucose positron-emission tomography/computed tomography for the postoperative surveillance of advanced renal cell carcinoma. BJU Int. 2009 Mar;103(5):615-9. doi: 10.1111/j.1464-410X.2008.08150.x. Epub 2008 Oct 24. PMID 19007371
- [Background] Majhail NS, Urbain JL, Albani JM, Kanvinde MH, Rice TW, Novick AC, Mekhail TM, Olencki TE, Elson P, Bukowski RM. F-18 fluorodeoxyglucose positron emission tomography in the evaluation of distant metastases from renal cell carcinoma. J Clin Oncol. 2003 Nov 1;21(21):3995-4000. doi: 10.1200/JCO.2003.04.073. PMID 14581422
- [Background] Lawrentschuk N, Davis ID, Bolton DM, Scott AM. Functional imaging of renal cell carcinoma. Nat Rev Urol. 2010 May;7(5):258-66. doi: 10.1038/nrurol.2010.40. PMID 20448659
- [Background] Sawicki LM, Buchbender C, Boos J, Giessing M, Ermert J, Antke C, Antoch G, Hautzel H. Diagnostic potential of PET/CT using a 68Ga-labelled prostate-specific membrane antigen ligand in whole-body staging of renal cell carcinoma: initial experience. Eur J Nucl Med Mol Imaging. 2017 Jan;44(1):102-107. doi: 10.1007/s00259-016-3360-2. Epub 2016 Mar 21. PMID 26996777
- [Background] Aide N, Cappele O, Bottet P, Bensadoun H, Regeasse A, Comoz F, Sobrio F, Bouvard G, Agostini D. Efficiency of [(18)F]FDG PET in characterising renal cancer and detecting distant metastases: a comparison with CT. Eur J Nucl Med Mol Imaging. 2003 Sep;30(9):1236-45. doi: 10.1007/s00259-003-1211-4. Epub 2003 Jul 4. PMID 12845486